CLINICAL TRIAL: NCT01649206
Title: Thyroid Nodules Treated With Percutaneous Radiofrequency Thermal Ablation: a Comparative Study
Brief Title: Percutaneous Radiofrequency Thermal Ablation in Compressive Thyroid Nodules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annamaria Colao, Department of Clinical and Molecular Endocrinology and Oncology, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTA-2012
Record Dates: First submitted 2012-07-16; First posted 2012-07-25 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Nodule; Radiofrequency Thermal Ablation; Pressure symptoms; Hyperthyroidism
MeSH Terms: conditions — Thyroid Nodule; Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: RTA (Experimental): Percutaneous Radiofrequency Thermal Ablation (RTA).
  Interventions: Procedure: Percutaneous Radiofrequency Thermal Ablation
- Group B: untreated (No Intervention): No treatment, only follow-up

INTERVENTIONS:
Procedure: Percutaneous Radiofrequency Thermal Ablation — Percutaneous Radiofrequency Thermal Ablation (RTA) by using a RITA© StarBurst Talon needle (RITA Medical Systems, Fremont, CA). RTA is performed in each patient at Time 0.
  Arms: Group A: RTA

SUMMARY:
Percutaneous radiofrequency thermal ablation (RTA) was reported as an effective tool for the management of thyroid nodules (TNs). This study aims to validate RTA as a valid approach for patients with compressive TNs for whom surgery is contraindicated or refused. Two groups of subjects with TNs (one group to treat with RTA and a matched untreated control group) will be evaluated in term of TN volume, thyroid hormones and clinical symptoms.

DETAILED DESCRIPTION:
Thyroid nodules (TNs) are very common in the general population, with a prevalence of about 50% in subjects older than 60 years undergoing neck ultrasound examination.

The great majority of TNs are benign, but they can be responsible for pressure symptoms in the neck and result in discomfort and decreased quality of life. Large compressive TNs may result in life-threatening conditions because of the potential acute onset of respiratory crisis. Percutaneous radiofrequency thermal ablation (RTA) is a minimally invasive procedure which has been firstly develop to treat patients with liver cancer and has been then used to treat both malignant and benign tumor nodules in many organs. RTA also represents a promising new approach for the management of TNs.The current prospective comparative study investigated the long-term effectiveness of RTA in patients with both toxic and non-toxic compressive TNs.

Forty consecutive patients with TNs with pressure symptoms were prospectively enrolled in this study. Patients were randomised as follows: 20 patients were treated with a single RTA session (group A) and 20 patients did not receive any treatment and were only followed-up (group B).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* benign thyroid nodules (TYR 2)
* solid or predominantly solid (colloid component < 30%) large (> 4.0 mL) thyroid nodules
* refusal and/or inefficacy of surgery and/or radioiodine therapy.

Exclusion Criteria:

* pregnancy
* malignant or suspicious thyroid nodules.

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TN volume | 12 months
  Evaluation of TN volume by using Ultrasonography.

SECONDARY OUTCOMES:
Efficacy on TN-related neck symptoms | From time to treatment until 12 months. Time point evaluations at 1, 3, 6, 12 months.
  Evaluation of TN-related neck symptoms scored separately as follows: 0 (absent), 1 (moderate), and 2 (severe). The sum of the individual scores generates a final score (SYS score) ranging from 0 to 6.
Efficacy on TN hyperfunction | Efficacy on TN-related neck symptoms Time Frame: (FDAAA) From time to treatment until 12 months. Time point evaluations at 1, 3, 6, 12 months.
  Evaluation of TN hyperfunction by measuring serum concentrations of TSH, free thyroxine (fT4), free triiodothyronine (fT3) in patients with toxic TNs.
Safety | At 1, 3, 6, 12 months after baseline.
  Assessment of local impairment (pain, oedema, skin damage). Assessment of thyroid dysfunction by measuring serum concentrations of fT3, fT4, TSH.
  Assessment of thyroid autoimmunity (anti-Thyroglobulin and anti-Thyroperoxidase antibodies).
Change from baseline in TN volume | 1 month
  Evaluation of TN volume by using Ultrasonography
Change from baseline in TN volume | 3 months
  Evaluation of TN volume by using Ultrasonography
Change from baseline in TN volume | 6 months
  Evaluation of TN volume by using Ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, Principal Investigator — "Federico II" University of Naples
Locations (1):
- "Federico II" University of Naples, Department of Clinical and Molecular Endocrinology and Oncology, Naples, Italy